CLINICAL TRIAL: NCT00317499
Title: Double-Blind, Randomized, Placebo-Controlled Study of Etanercept (ENBREL) in the Treatment of Psoriatic Arthritis (PsA) and Psoriasis
Brief Title: Double-blind, Randomized, Placebo-controlled Phase 3 Study of Etanercept in the Treatment of Psoriatic Arthritis and Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20021630
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Psoriatic Arthritis; Psoriasis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Etanercept (Experimental)
  Interventions: Drug: Etanercept
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo
  Arms: Placebo
Drug: Etanercept — Etanercept
  Arms: Etanercept

SUMMARY:
This was a phase 3, double-blind, placebo-controlled, randomized, multicenter study in subjects with psoriatic arthritis (PsA) and psoriasis comprising 3 periods: a 24-week double-blind period, a ≤ 24-week maintenance period, and a 48-week open-label period. During the double-blind period, subjects were randomized equally to 1 of 2 regimens: etanercept 25 mg twice weekly (BIW) or placebo, administered subcutaneously (SC). After the week 24 visit, subjects continued on blind-labeled therapy in a maintenance period until all subjects completed the double-blind period. After the maintenance period, all subjects received open-label etanercept 25 mg BIW.

DETAILED DESCRIPTION:
Previously presented data from 2 double-blind, placebo-controlled trials (Protocols 016.0612 [Investigator IND] and 016.0030 [Immunex IND]) led to the approval of etanercept for reducing clinical signs and symptoms of PsA. One-year radiographic data from Protocol 20021630 led to an additional approval of etanercept for inhibiting structural progression in PsA.

Data are used for the following purposes:

* To summarize the clinical efficacy and safety results previously described in the 6-month clinical study report and the radiographic results previously described in the 1-year clinical study report.
* To show the effect of etanercept on physical function in subjects with PsA and psoriasis, as measured by 2 patient-reported outcome measures (disability index of the Stanford Health Assessment Questionnaire [HAQ] and Medical Outcomes Study Short-form Health Survey [SF-36]). • To present the radiographic results at 2 years from baseline and the final clinical efficacy and safety results during the open-label period of the study.

ELIGIBILITY:
Inclusion Criteria: Subjects had to satisfy the following criteria before randomization into the study:

* Active PsA at the time of screening, including ≥ 3 swollen joints and ≥ 3 tender/painful joints. • Had ≥ 1 of the following subtypes of PsA: distal interphalangeal (DIP) involvement; polyarticular arthritis (absence of rheumatoid nodules and presence of psoriasis); arthritis mutilans; asymmetric peripheral arthritis; or ankylosing spondylitis-like.
* Arthritis had demonstrated an inadequate response to nonsteroidal antiinflammatory drug (NSAID) therapy.
* Subjects had plaque psoriasis with qualifying target lesion. Target lesion was to be ≥ 2 cm in diameter and could not be on the scalp, axilla, or groin. Psoriasis was to be stable (ie, not accelerating).
* Between 18 and 70 years of age.
* Subjects remaining on concomitant MTX (≤ 25 mg/week) had inadequate disease control in the opinion of the investigator and had been on a stable dose of MTX for 2 months before start of investigational product. Subjects were required to maintain a stable dose of MTX throughout the study.
* Negative serum pregnancy test within 14 days before the first dose of investigational product in all women (except those surgically sterile or ≥ 5 years postmenopausal).
* Heterosexually active men and women of childbearing potential agreed to use a medically accepted form of contraception throughout the study, including the exclusionary medicine washout period and follow-up period.
* Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2 times laboratory's upper limit of normal; hemoglobin ≥ 8.5 g/dL; platelet count ≥ 125,000/mm3; white blood cell count ≥ 3,500 cells/mm3; and serum creatinine ≤ 2 mg/dL.
* Negative HIV test. Negative test for hepatitis B surface antigen and hepatitis C.
* Able to reconstitute and self-inject investigational product or have a designee who could do so.
* Capable of understanding and giving written, voluntary informed consent.

Exclusion Criteria:

* Guttate or pustular psoriasis.
* Evidence of skin conditions (eg, eczema) other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis.
* Active severe infection within 1 month of investigational product administration.
* Subjects must be off antibiotics for 1 week before investigational product administration.
* Previous receipt of etanercept, known antibody to TNF, or experimental metalloproteinase inhibitors (past or current use of minocycline and doxycycline was acceptable).
* Receipt of investigational drugs or biologics within 4 weeks of the screening visit.
* Receipt of anti-CD4 or diptheria IL-2 fusion protein within the previous 6 months, with a subsequent abnormal absolute T cell count.
* Psoralen ultraviolet A phototherapy (PUVA) within 4 weeks of investigational product initiation. Ultraviolet B (UVB) phototherapy within 2 weeks of investigational product initiation.
* Receipt of disease-modifying anti-rheumatic drugs (DMARDs) other than MTX (eg, hydroxycholorquine, oral or injectable gold, cyclophosphamide, cyclosporine, azathioprine, D-penicillamine, or sulfasalazine) or intra-articular corticosteroids within 4 weeks before the first dose of investigational product.
* Dose of NSAID greater than the maximum recommended dose in the product information. NSAID dose had to be stable for ≥ 4 weeks before screening evaluation.
* Concomitant corticosteroids > 10 mg/day of prednisone (or its equivalent). Corticosteroid dose had to be stable for ≥ 4 weeks before screening evaluation.
* Topical steroids, oral retinoids, topical vitamin A or D analog preparations or anthralin within 14 days of baseline. (Exception: Topical therapies were permitted on scalp, axillae, and groin but had to be stable throughout trial.)
* Pregnancy or lactation in women.
* Significant concurrent medical diseases including:

  * Diabetes mellitus requiring insulin
  * Uncompensated congestive heart failure
  * Myocardial infarction within 12 months of screening visit
  * Unstable or stable angina pectoris
  * Uncontrolled hypertension
  * Severe pulmonary disease (requiring medical or oxygen therapy)
  * History of cancer (other than resected cutaneous basal or squamous cell carcinoma or in situ cervical cancer) within 5 years of screening visit
  * HIV positive, hepatitis B surface antigen, or hepatitis C positive
  * Rheumatoid arthritis, systemic lupus, scleroderma, or polymyositis
  * Any condition judged by the subject's physician that would cause this study to be detrimental to the subject
* Current or history of psychiatric disease that would interfere with ability to comply with the study protocol or give informed consent.
* History of alcohol or drug abuse that would interfere with ability to comply with the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2000-04; Primary Completion 2002-06 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Mease PJ, Ritchlin CT, Martin RW, Gottlieb AB, Baumgartner SW, Burge DJ, Whitmore JB. Pneumococcal vaccine response in psoriatic arthritis patients during treatment with etanercept. J Rheumatol. 2004 Jul;31(7):1356-61. PMID 15229957
- [Result] Mease PJ, Kivitz AJ, Burch FX, Siegel EL, Cohen SB, Ory P, Salonen D, Rubenstein J, Sharp JT, Tsuji W. Etanercept treatment of psoriatic arthritis: safety, efficacy, and effect on disease progression. Arthritis Rheum. 2004 Jul;50(7):2264-72. doi: 10.1002/art.20335. PMID 15248226
- [Result] Mease PJ, Kivitz AJ, Burch FX, Siegel EL, Cohen SB, Ory P, Salonen D, Rubenstein J, Sharp JT, Dunn M, Tsuji W. Continued inhibition of radiographic progression in patients with psoriatic arthritis following 2 years of treatment with etanercept. J Rheumatol. 2006 Apr;33(4):712-21. Epub 2006 Feb 1. PMID 16463435
- [Result] Bansback NJ, Ara R, Barkham N, Brennan A, Fraser AD, Conway P, Reynolds A, Emery P. Estimating the cost and health status consequences of treatment with TNF antagonists in patients with psoriatic arthritis. Rheumatology (Oxford). 2006 Aug;45(8):1029-38. doi: 10.1093/rheumatology/kel147. Epub 2006 Jun 16. PMID 16782734
- [Result] Mease PJ, Woolley JM, Singh A, Tsuji W, Dunn M, Chiou CF. Patient-reported outcomes in a randomized trial of etanercept in psoriatic arthritis. J Rheumatol. 2010 Jun;37(6):1221-7. doi: 10.3899/jrheum.091093. Epub 2010 Apr 15. PMID 20395648
- [Derived] Mease PJ, Woolley JM, Bitman B, Wang BC, Globe DR, Singh A. Minimally important difference of Health Assessment Questionnaire in psoriatic arthritis: relating thresholds of improvement in functional ability to patient-rated importance and satisfaction. J Rheumatol. 2011 Nov;38(11):2461-5. doi: 10.3899/jrheum.110546. Epub 2011 Sep 1. PMID 21885498
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com